CLINICAL TRIAL: NCT01522300
Title: Etude Tomos- Apport de la Tomosynthèse Dans le Bilan d'Extension locorégional préthérapeutique d'Une Tumeur du Sein : Recherche de multicentricité
Brief Title: Etude Tomos- Apport de la Tomosynthèse Dans le Bilan d'Extension locorégional préthérapeutique d'Une Tumeur du Sein : Recherche de multicentricité Tomos Study- Contribution of Tomosynthesis In Locoregional Pretherapeutic Staging of a Breast Tumor: Multicentricity Search
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No more inclusions since august 2013
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TOMOS
Record Dates: First submitted 2012-01-18; First posted 2012-01-31 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Mammary Tumor
Keywords: Tomosynthesis; breast cancer; specificity; sensitivity; To assess efficacy of Tomosynthesis by evaluating its sensitivity and specificity in detecting the multicentricity of mammary tumor
MeSH Terms: conditions — Breast Neoplasms; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Evaluation of the Tomosynthesis — An exam by tomosynthesis will be realised at the inclusion of the patient in the study.
Other: Avaluation of a medical device: the tomosynthesis — An exam by tomosynthesis will be realised at the inclusion of the patient in the study

SUMMARY:
The main objective of the study is to assess the sensitivity and specificity of Tomosynthesis in detecting the multicentricity of mammary tumor.

DETAILED DESCRIPTION:
The secondaries objectives of the study are:

* Sensitivity and specificity in detecting multifocality of breast tumor
* Sensitivity and specificity of Tomosynthesis in the detection of contralateral tumors
* Predetermination of potential targets for ultrasound

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years.
* Patients with a breast tumor, regardless of the stage and size
* Compulsory affiliation to a social security system.
* Obtaining informed consent in writing, signed and dated.

Exclusion Criteria:

* Patients with cognitive or psychiatric disorders.
* Patient deprived of liberty by a court or administrative.
* Patients with indications against the achievement of MRI, mammography and tomosynthesis
* Pregnant Women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To calculate the sensitivity and specificity of both types of imaging (mammography and Tomosynthesis) with respect to number of tumors multicentric and multifocal identified through MRI. | January 2013
  To calculate the sensitivity and specificity of both types of imaging (mammography and Tomosynthesis) with respect to number of tumors multicentric and multifocal identified through MRI. The other parameters VPN, VPP will also be calculated and discussed.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Jean Perrin, Clermont-Ferrand, France